CLINICAL TRIAL: NCT07245238
Title: Efficacy of Topical Cannabidiol Lotion for Pruritus Relief, Hydrating, Sleep Quality, Quality of Life Improvement in Systemic Sclerosis: a Randomized Double Blinded Controlled Crossover Trial
Brief Title: Topical Cannabidiol Lotion for Pruritus Relief in Scleroderma
Acronym: cannabidiol
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Chingching Foocharoen, Principle investigator, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cannabidiol cream; Khon Kaen University (Other Grant/Funding Number: Khon Kaen University)
Record Dates: First submitted 2025-11-15; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Mediciine; Systemic Sclerosis (SSc); Intervention Study
Keywords: systemic sclerosis; Cannabinoid; Emollients; Crossover study design; Randomized controlled trial; Sleep quality; Pruritus; \Cannabidiol; Cannabidiol
MeSH Terms: conditions — Scleroderma, Systemic; Sleep Initiation and Maintenance Disorders; Pruritus | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): 10% urea lotion
  Interventions: Drug: Control
- Treatment (Experimental): 10% urea lotion plus 1% cannabidiol
  Interventions: Drug: 10% urea lotion plus 1% cannabidiol

INTERVENTIONS:
Drug: 10% urea lotion plus 1% cannabidiol — 10% urea lotion plus 1% cannabidiol
  Arms: Treatment
Drug: Control — 10% urea lotion
  Arms: Control

SUMMARY:
Itching is one of the common symptoms found in patients with scleroderma, with a prevalence of about 42-62%, and it often occurs in the early stages of the disease. The mechanisms of itching are still unclear, and current treatments have not yet shown any clear efficacy in alleviating itching caused by scleroderma. Hemp extract has previously been used to treat itching in chronic skin diseases. Besides its antipruritic (anti-itch) effect, hemp extract also possesses anti-inflammatory properties, increases skin moisture, and helps repair the skin, all without psychoactive effects.

Studies have investigated the benefits of hemp extract in the form of a topical cream with concentrations ranging from 1-5% for the treatment of various skin diseases such as psoriasis, eczema, and the management of fingertip ulcers in scleroderma patients. The results showed that a 1% hemp extract cream relieved itching in eczema and at the same concentration also helped heal fingertip ulcers in scleroderma patients. However, to date, there has been no clear study on the effectiveness of hemp extract in cream or lotion form for treating itching in scleroderma patients. Additionally, there is currently no standard guideline for the management of itching in scleroderma. Generally, 10% urea cream is commonly used to increase skin moisture and alleviate itching, but there has been no prior study on its efficacy specifically for itch relief.

Therefore, this study aims to evaluate the efficacy of a 1% hemp extract combined with 10% urea in lotion form compared to a lotion containing only 10% urea (without hemp extract) in relieving itching, increasing skin moisture, and reducing sleep disturbances caused by itching in scleroderma patients, as well as assessing any potential side effects.

DETAILED DESCRIPTION:
Systemic Sclerosis (SSc), also known as scleroderma, is a connective tissue disease primarily characterized by skin hardening. It can be classified into two main subgroups: limited cutaneous systemic sclerosis (lcSSc) and diffuse cutaneous systemic sclerosis (dcSSc), based on the extent of skin involvement.

Currently, there are no definitive studies on the efficacy of topical Cannabidiol (CBD) for treating pruritus in SSc patients. Furthermore, there is no standardized guideline for the management of pruritus in SSc in general. A 10% urea cream is commonly used to improve skin hydration and reduce itching.

This study aims to evaluate the efficacy of a lotion containing 10% urea combined with 1% CBD, formulated for ease of administration and a comfortable, non-greasy feel. This formulation will be compared against a lotion containing only 10% urea. The study will assess its effectiveness in relieving pruritus, improving skin hydration, and reducing sleep disturbances caused by itching in patients with systemic sclerosis. It will also evaluate any potential side effects.

Primary Objective

To compare the efficacy of a 10% urea lotion with 1% topical CBD (investigational group) versus a 10% urea lotion alone (control group) in alleviating pruritus in patients with systemic sclerosis.

Secondary Objectives

To compare the effects of the investigational and control groups on skin hydration.

To compare the effects of the investigational and control groups on skin melanin levels and erythema (redness).

To compare the effects of the investigational and control groups on sleep quality.

To compare the effects of the investigational and control groups on quality of life.

To assess the change in pruritus from baseline after two weeks of treatment. To evaluate adverse events associated with the use of the investigational and control products.

ELIGIBILITY:
Inclusion Criteria:

1. SSc patients aged between 18 and 70 years
2. Diagnosed according to ACR/EULAR 2013 classification criteria
3. Having chronic pruritus
4. Must not receive steroid equivalent to prednisolone dose more than 10 mg/d
5. Must receive a stable dose of steroid, immunosuppressant and/or vitamin or its supplement within 2 weeks before enrollment
6. Must stop moisturizer treatment at least 1 week prior to randomization
7. Must stop anxiolytics, hypnotics or sleeping pills at least 2 weeks before enrollment
8. Understand and able to read and write Thai language

Exclusion Criteria:

1. Overlap with other connective tissue diseases
2. Pregnancy or lactation
3. Bedridden and confined to no self-care
4. Evidence of active malignant disease
5. Present of uncontrolled or severe medical problems including diabetes mellitus, asthma, angina, cardiovascular, thyroid, hepatobiliary included cholestasis, or renal diseases (Cr>1.4 mg/dl)
6. Present of active infection that needs systemic antibiotic
7. Previous allergy to urea cream, cannabinoid or its derivatives
8. Concomitant illegal drug used (amphetamine or its derivative, cocaine)
9. On-going anxiolytics, hypnotics or sleeping pills used
10. In a period that needs immunosuppressant dose adjustment
11. Having history of schizophrenia, concurrent active mood disorder, or anxiety disorders
12. Having dermatologic diseases causing pruritus such as atopic dermatitis, contact dermatitis, psoriasis, folliculitis, urticaria, lichen planus, bullous pemphigoid, dermatophytosis, pediculosis, scabies, cutaneous T cell lymphoma, sunburn, drug allergy or skin eruption
13. Having systemic diseases causing of pruritus other than SSc such as neurologic disease, polycythemia vera

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The changing of intensity of pruritus evaluated by visual analogue scale (VAS) compared to baseline and a comparison between treatment and control group | 2 weeks
  The changing of intensity of pruritus evaluated by visual analogue scale (VAS) compared to baseline and a comparison between treatment and control group

SECONDARY OUTCOMES:
The changing of course of pruritus evaluated by Dynamic Pruritus Score compared to baseline in each group | 2 weeks
  The changing of course of pruritus evaluated by Dynamic Pruritus Score compared to baseline in each group
The changing of skin hydration evaluated by using the Corneometer CM 825 compared to baseline and a comparison between treatment and control at the same skin area | 2 weeks
  The changing of skin hydration evaluated by using the Corneometer CM 825 compared to baseline and a comparison between treatment and control at the same skin area
The changing of skin melanin content and erythema level evaluated by using the Mexameter MX 18 compared to baseline and a comparison between treatment and control at the same skin area | 2 weeks
  The changing of skin melanin content and erythema level evaluated by using the Mexameter MX 18 compared to baseline and a comparison between treatment and control at the same skin area
The changing of course of pruritus evaluated by Patient Benefit Index compared to baseline in each group | 2 weeks
  The changing of course of pruritus evaluated by Patient Benefit Index compared to baseline in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided